CLINICAL TRIAL: NCT06812845
Title: Patterns of Eye Diseases Among Patients Attending The Eye Investigation Unit of Sohag University Hospital
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mahmoud Abd Elwareth Mohamed, mahmoud abd elwareth, Sohag University
Other Study IDs: Soh-Med--25-1-10MS
Record Dates: First submitted 2025-02-01; First posted 2025-02-06 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Eye Diseases
Keywords: patterns of eye disease
MeSH Terms: conditions — Eye Diseases | interventions — Visual Acuity; Refraction, Ocular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: eye investigations — BY data entry ,measuring the visual acuity ,measuring IOP, doing refraction and recording eye investigations results to reach the final diagnosis
  Other Names: visual acuity; IOP measurment; Refraction

SUMMARY:
The goal of the work: is to assess the patterns of eye diseases in patients attending the eye investigation unit of Sohag University Hospital.organize the community education. The main question it aims to answer is

* DOES eye disease blindness prevalence rate increase in women more than men?
* What is the rate of glaucoma and other ocular diseases that causes irreversible blindness among the attending patients? Patients attending to the eye investigation unit of Sohag University Hospital in the period from January 2025 to December 2025 are being observed in this work to determine the eye diseases prevalence.

DETAILED DESCRIPTION:
This type of study is helpful to get an idea about the epidemiology of ocular disorders. It is necessary to organize the community education and ensure early treatment to reduce the prevalence of such diseases in the general population.

* Aim of the work: is to assess the patterns of eye diseases in patients attending the eye investigation unit of Sohag University Hospital.
* Study design: observational Cross-Sectional study.3
* Patients and methods: all patients attending to the eye investigation unit of Sohag University Hospital in the period from January 2025 to December 2025.
* Inclusion criteria: All patients referred to the eye investigation unit from the outpatient clinic of Sohag university hospital, private clinics or health insurance.
* Exclusion criteria:

  1. Patients unable to measure visual acuity.
  2. Patients unable to measure intraocular pressure.
  3. Mentally retarded patients.
  4. Undiagnosed patients.
* Time schedule:

  1. Twelve months for collection of data, writing the review of literature and methodology.
  2. Three months for analysis of data and writing the results.
  3. Three months for writing the discussion and conclusions.
* ethical considerations:

  1. The study adheres to Tents of Helsinki declaration.
  2. The study will be approved by the ethical committee of the faculty of medicine Sohag University.
  3. An informed written consent will be taken from all of the participants in the study or their guardians

ELIGIBILITY:
Inclusion Criteria:

- All patients referred to the eye investigation unit from the outpatient clinic of Sohag university hospital, private clinics or health insurance.

Exclusion Criteria:

* Patients unable to measure visual acuity.
* Patients unable to measure intraocular pressure.
* Mentally retarded patients.
* Undiagnosed patients.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: all patients attending to the eye investigation unit of Sohag University Hospital in the period from January 2025 to December 2025.
Sampling Method: Non-Probability Sample
Enrollment: 7000 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
determine the pattrens of eye diseases among patients attending the eye investigtion unit of sohag university | 1. Twelve months for collection of data, writing the review of literature and methodology. 2. Three months for analysis of data and writing the results. 3. Three months for writing the discussion and conclusions.
  recording data of the prevalence of each eye disease among the study group in the period from January 2025 to December 2025 .their percentage in men and women , also in which age group

CONTACTS AND LOCATIONS:
Overall Officials: mortada AH Prof\ abuzaid, Professor, Study Director — depatement of ophthalmology ,sohag university
Locations (1):
- Faculty of Medicine in Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided